CLINICAL TRIAL: NCT06378229
Title: Psilocybin-assisted Psychotherapy in the Treatment of Patients Hospitalized for Treatment-resistant Depression: an Open-label Feasibility Study with an Experiential and Systemic Focus
Brief Title: Psilocybin for Hospitalized Patients with Treatment-resistant Depression
Acronym: PSIHOS-D
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Filament Health Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0157; 2022-501857-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-14; First posted 2024-04-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Open label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label: full dose Psilocybin (Experimental): 2 doses of 25mg Psilocybin, 3 weeks apart (week 3 and week 6), accompanied by 7,5 hours of preparation sessions and 9 hours of integration sessions.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — A psychedelic drug found in certain mushrooms. It will be in a capsule of 25mg psilocybin (PEX010).
  Other Names: PEX010

SUMMARY:
The purpose of this study is to determine the safety and feasibility of performing psilocybin-assisted psychotherapy in patients hospitalized for treatment-resistant depression.

DETAILED DESCRIPTION:
The proposed study will assess the safety, feasibility, preliminary results and neurological aspects of psilocybin-assisted psychotherapy in the treatment of hospitalized patients with treatment-resistant depression.

Screening, after signing the ICF, is done in patients newly admitted to the psychiatric service of Ghent University Hospital or patients referred for hospitalization through the outpatient clinic of the psychiatric service of Ghent University Hospital. Involved patients are hospitalized at the Anxiety, Compulsion and Mood Unit for 8 weeks. They will receive add-on treatment with psilocybin-supported psychotherapy in addition to standard treatment (daily group therapies, mainly non-verbal and activating). This consists of a preparatory phase (4 sessions of 1.5 hours before the first psilocybin session and 1 session of 1.5 hours before the second psilocybin session), the psilocybin sessions themselves (2 sessions, week 3 and week 6) and an integration phase (3 sessions of 1.5 hours after each psilocybin session). All sessions occur with the same 2 therapists throughout the entire course. Therapists are trained to provide experiential and systemic psychotherapeutic interventions.

After hospitalization, weekly outpatient follow-up consultations continue until 12 weeks after the last psilocybin session. Subsequently, patients may still agree to a prospective, observational and naturalistic follow-up until 1 year after the last psilocybin session, during which they will be called monthly by a psychiatrist from the research team to inquire about current mental status and any therapies undertaken in the interim.

During the study, patients are required to fill out questionnaires at regular intervals. Video-recordings will be made of certain parts of the preparation and integration sessions, for analysis with the client experience scale (EXP). The morning of each psilocybin session, female patients must provide a blood sample for a pregnancy test. The morning of each psilocybin session, all patients must provide a urine sample for toxicology screening. EEGs are also taken from patients the day before each psilocybin session, the morning of the first integration session after each psilocybin session and 12 weeks after the last psilocybin session (at the last outpatient consultation). At the start and at the end of the hospitalization phase, a semi-structured interview will be conducted with the patient to gauge expectations on the one hand and experiences on the other.

Throughout the study, the patient's partner will be involved. The partner must complete a number of questionnaires at baseline and throughout the study and will have to be present at 3 EEGs. In addition, the partner will also participate in 1 preparatory session and 2 integration sessions. The partner will also be given the opportunity to spend the night of a psilocybin session with the patient in the hospital (rooming-in). At the start and at the end of the hospitalization phase, a semi-structured interview will be conducted with the partner to gauge expectations on the one hand and experiences on the other.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of major depressive disorder (single and recurrent episodes) of moderate to severe degree (MADRS score ≥ 20) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), without psychotic features. Included ICD-11 diagnoses are ICD-11: 6A70.1, 6A70.3, 6A71.1, 6A71.3.
3. Subjects have failed to respond to 2 or more antidepressants prescribed at the minimum effective dose for at least 6 weeks. Augmentation with an add-on treatment counts as a second treatment.
4. The subjects are abstinent from alcohol (breathalyzer blood alcohol concentration (BAC) level 0.00) and provide a negative urine drug screen at the dosing day.
5. The female subjects provide a negative pregnancy test at the dosing day.
6. The subjects must be medically stable based on clinical laboratory tests, medical history, vital signs, and 12-lead ECG performed at screening.

   - In 12-lead ECG, QTcF should be ≤ 450 ms for males or ≤ 470 ms for females and PR-interval < 220 ms at screening.
7. A partner is willing to participate in the study (a cohabiting relationship of at least 1 year).

Exclusion Criteria:

1. Currently comorbid or previously diagnosed DSM-5 diagnosis of a

   1. major depressive episode with psychotic features.
   2. psychotic disorder (defined as meeting DSM-5 criteria for any psychotic disorder) on the MINI 7.0, EXCEPT substance/medication induced psychotic disorder where the duration was limited to the acute period of direct intoxication with the substance/medication. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
   3. bipolar disorder (defined as meeting DSM-5 criteria for bipolar type 1 or bipolar type 2) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
   4. drug or alcohol dependence syndrome (defined as meeting DSM-5 criteria for any dependence syndrome) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
   5. cluster B personality disorder. Subjects will be screened for the presence of those personality traits by using the NEO-FFI-3.
   6. PTSD (defined as meeting DSM-5 criteria for PTSD) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
2. A family history (first-degree relative) of psychosis and/or bipolar disorder.
3. Current active suicidal ideations.
4. Depression secondary to other medical conditions.
5. Medical diagnosis incompatible with psilocybin treatment:

   1. Cardiovascular conditions: recent stroke (< 1 year from signing of ICF), recent myocardial infarction (< 1 year from signing of ICF), uncontrolled hypertension (blood pressure > 140/90 mmHg) or clinically significant arrhythmia within 1 year of signing the ICF.
   2. Uncontrolled insulin-dependent diabetes mellitus.
   3. Uncontrolled epilepsy.
6. Biochemical or electrocardiographic abnormalities determined as clinically significant by a medical doctor. PsiHos-D, Version 2.1 dd. 22/02/2024 page 59 of 114 TMP_Protocol AGO CTR_Version 1.0_Effective Date 2022-07-18
7. Current intake of Lithium, Disulfiram, MAOIs or inhibitors of UGT1A9 and 1A10.
8. The subject has received any prior treatment with vagal nerve stimulation, or a deep brain stimulation device.
9. Women of childbearing potential not using adequate contraception (methods that can achieve a failure rate of less than 1%: combined hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence). A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
10. Pregnant or breast-feeding women.
11. Those unable to give informed consent.
12. Those enrolled in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of Treatment-Emergent Adverse Events | 18 weeks
  The safety of performing psilocybin-assisted psychotherapy in treatment-resistant depression (TRD) in a hospitalized setting. Adverse Events (AEs) will be classified by the clinical team based on severity, whether they are expected or unexpected and causality.
Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 weeks
  Clinician-administered measure of suicidal ideation. Scores range from 0 to 25, with higher scores indicating more severe suicidal ideation.

SECONDARY OUTCOMES:
Recruitment and retention rates. | 8 weeks (end of hospitalization).
  The feasibility of performing psilocybin-assisted psychotherapy in TRD in a hospitalized setting.
Qualitative data from the semi-structured interviews with the subjects and their partners. | 8 weeks (end of hospitalization).
  Acceptability of the intervention and procedures for the subjects as assessed through semi-structured interviews.

OTHER OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 18 weeks (optional up to 58 weeks).
  A ten-item clinician-rated diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Scoring ranging from 0 to 60, with higher scores indicating greater depressive symptomology.
Quick Inventory of Depressive Symptomatology - Self Rated (QIDS-SR) | 18 weeks.
  A self report measure of depressive symptoms. Scores range from 0 to 27, with lower scores indicating less symptoms of depression.
State-Trait Anxiety Inventory (STAI) | 18 weeks.
  A self report measure of anxiety symptoms. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
World Health Organization Quality of Life Inventory-Brief subscale (WHOQOL-BREF) | 18 weeks (optional up to 58 weeks).
  A self-report measure of quality of life with four subscales: Physical Health, Psychological Health, Social Relationships, and Environment. Scores for each range from 4-20, with higher scores indicating better quality of life.
Maudsley 3-item Visual Analogue Scale (M3VAS) | 18 weeks.
  A self report measure of depressive symptoms using 3 visual analogue scales. Scores range from 0 to 300, with lower scores indicating less symptoms of depression.
Subjective Emotional Health Visual Analogue Scale (SEHVAS) | 18 weeks.
  Visual Analogue Scale rating the emotional health of the subject as perceived by the partner. Scores range from 0 to 100, with higher scores indicating a better emotional health.
revised Dyadic Adjustment Scale (RDAS) | 18 weeks (optional up to 58 weeks).
  A 14-item questionnaire that measures an individual's perceptions of his/her relationship with an intimate partner. Scores range from 0-69, with higher scores indicating higher consensus, satisfaction and cohesion.
Zarit Burden Interview - Short Form (Zarit-12 Burden Scale) | 18 weeks.
  A self-administered 12-item questionnaire that measures the burden of taking care for a close relative. Scores range from 0 to 48, with higher scores indicating a greater burden of care.
Client Experiencing Scale (EXP) | Week 2, 3, 5 and 6.
  A 7-item scale assessing the experiential level of the subject. Higher stages indicate higher levels of experiencing.
Mystical Experience Questionnaire (MEQ) | Within 24 hours after each psilocybin session (week 3 and week 6).
  A 30-item questionnaire that measures the mystical quality of an experience. Scores range from 0 to 5, with higher scores indicating a greater mystical quality of the experience.
Working Alliance Inventory - Short Revised (WAI-SR) | 8 weeks.
  A 12-item questionnaire that measures the quality of the therapeutic relationship. Scores range from 1 to 5, with higher scores indicating better quality of the therapeutic relationship.
Semi-structured interviews. | Week 1 and week 8.
  Semi-structured interviews with both subjects and their partners, assessing their expectations and experiences.
EEG: sensor level analysis (power) and source level analysis (functional connectivity through amplitude envelope correlation), both in resting state and during an emotional paradigm. | Week 3, week 6, week 18.
  A method aimed at examining intrinsic networks in the brain to estimate correlations between brain regions.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Lemmens, Prof. dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF